CLINICAL TRIAL: NCT02481674
Title: A Phase 2, Multi-center, Randomized, Double-blind, Placebo Controlled Study in Subjects With Late Prodromal and Early Manifest Huntington's Disease to Assess the Safety, Tolerability, pk, and Efficacy of Pepinemab
Brief Title: A Study in Subjects With Late Prodromal & Early Manifest HD to Assess the Safety, Tolerability, pk, and Efficacy of Pepi
Acronym: SIGNAL-HD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vaccinex Inc. (Industry)
Collaborators: Huntington Study Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX15/2503-N-131
Record Dates: First submitted 2015-06-19; First posted 2015-06-25 (Estimated); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Huntington's Disease
Keywords: Prodromal Stage; Early Manifest Stage
MeSH Terms: conditions — Huntington Disease; Prodromal Symptoms | interventions — pepinemab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VX15/2503 (Experimental): The study drug VX15/2503 will be administered via monthly intravenous infusions
  Interventions: Drug: VX15/2503
- Placebo (Placebo Comparator): A placebo control will be administered via monthly intravenous infusions
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VX15/2503 — VX15/2503 (pepinemab) is a humanized IgG4 monoclonal antibody and will be administered intravenously at a dose of 20 mg/kg. The antibody is formulated at 20 mg/mL in 20 mM Sodium Acetate buffer, pH 5.4, containing 130 mM Sodium Chloride and 0.02% Polysorbate 80.
  Other Names: pepinemab
  Arms: VX15/2503
Drug: Placebo — Placebo consists of formulation buffer only which is 20 mM Sodium Acetate buffer, pH 5.4, containing 130 mM Sodium Chloride and 0.02% Polysorbate 80.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, PK, and efficacy of Pepinemab in subjects with late prodromal and early manifest Huntington's disease.

DETAILED DESCRIPTION:
VX15/2503-N-131 (SIGNAL-HD) is a Phase 2, multi-center, randomized, double-blind, placebo controlled study of VX15/2503 (pepinemab) in subjects with late prodromal and early manifest Huntington's disease. The primary objective is to evaluate the safety and tolerability of monthly IV administration of a single dosage of pepinemab (or placebo). Efficacy endpoints include determining the effect of pepinemab on brain volumes (MRI), FDG-PET imaging, 11C-PBR28 (TSPO) PET imaging (subset of Cohort B only) and clinical features of HD including cognition, motor function, behavior, functional abilities, global function and global measurement of change. Additional endpoints include PK / PD, immunogenicity, and exploratory biomarkers. Subjects in Cohort B that have received 12 months of pepinemab who volunteer will undergo a lumbar puncture at V13 to collect cerebral spinal fluid (CSF) to evaluate pepinemab mAb concentrations, total sSEMA4D levels, and other biomarkers in their CSF. Enrollment will involve approximately 276 individuals who are 21 years of age or older with late prodromal (CAG-age product score (CAP score) of greater than 200 and Diagnostic Confidence Level (DCL) of 2 or 3) or early manifest HD (Total Functional Capacity (TFC) greater than or equal to 11). The study will be divided into Cohort A and Cohort B. Cohort A is now complete and an unblinded analysis has been performed. Cohort A subjects were treated for 6 months with either drug or placebo (1:1) and then all subjects were treated with drug for 6 months, followed by 3 months of follow up. Treatment duration for each subject in Cohort A was 12 months. Participation in Cohort A included a Screening visit, a Baseline visit within 30 days of screening; 12 monthly treatment visits beginning at baseline and continuing through Month 12; follow-up safety phone call at one month and a follow-up safety visit three months after the final infusion. Cohort A subjects participated in the study for approximately 16 months. Based on the analysis of Cohort A, it was decided to extend the duration of treatment for a subset of subjects in Cohort B to evaluate the clinical response to pepinemab after 36 months. Additional enrolled subjects in Cohort B will be treated with drug or placebo (1:1). Participation in Cohort B will include a Screening visit, a Baseline visit within 30 days of screening; 18 or 36 monthly visits beginning at baseline and continuing through Month 18 or Month 36; follow-up safety phone call or visit, and for a subset of subjects, a follow-up safety visit three and six months after the final infusion. Cohort B subjects will participate in the study for approximately 19 and up to 37 months.

ELIGIBILITY:
Inclusion Criteria Highlights:

1. Male or female and are at least greater than or equal to 21 years of age at Screening.
2. Must fulfill one of the following criteria at Screening:

   1. Late prodromal HD as defined by a CAP score of greater than 200 and DCL 2 or 3.
   2. Early manifest HD as defined by a TFC greater than or equal to 11. Subject must have been determined to have a clinical diagnosis of HD by the Site Investigator as defined by a DCL of 4.
3. Must fulfill both of the following criteria at Screening:

   1. Have undergone genetic testing with a known CAG repeat greater than or equal to 36.
   2. No features of juvenile HD (Westphal variant).
4. If female must be either surgically sterile, postmenopausal, or nonlactating and nonpregnant. Female subjects of childbearing potential must practice a highly effective method of contraception.
5. If male, must agree to use a reliable method of birth control (condoms with contraceptive foams or sexual abstinence) during the study and for 6 months after the last dose of study drug.
6. Are willing and capable of providing informed consent for study participation, CAG genotyping (all subjects).
7. Are capable of reading, writing, and communicating effectively with others.
8. Are taking stable doses of any concomitant medications (including tetrabenazine and deutetrabenazine) during the 1 month prior to the Baseline Visit, with the exception of newly prescribed anxiolytics for the use of pre-medication prior to imaging at screening, which will be permitted on a case-by-case basis.
9. Must meet all criteria required to move forward with the Randomization Authorization Flow (RAF) and be considered eligible by the RAF Reviewer.

Exclusion Criteria Highlights:

1. Have participated in an investigational drug or device study within 30 days of the Baseline Visit, or 180 days if previous investigational drug was a MAb therapeutic, or previously participated in SIGNAL Cohort A. This does not apply to Cohort B subjects who are being offered the option to participate in the extension of Cohort B.
2. Have had previous neurosurgery for Huntington's disease or other movement disorders.
3. Are a suicide risk, as determined by meeting any of the following criteria:

   1. suicide attempt within one year prior to Baseline.
   2. suicidal ideation as defined by a positive response to question 5 on the C-SSRS (Baseline visit form) suicidal ideation section, within 60 days of the Baseline Visit.
   3. significant risk of suicide, as judged by the site Investigator.
4. Have marked cognitive impairment with a Montreal Cognitive Assessment (MoCA) Score less than or equal to 22.
5. Have a presence of clinically significant psychosis and/or confusional states, in the opinion of the site Investigator.
6. Have clinically significant laboratory or ECG abnormalities at Screening, in the opinion of the site Investigator.
7. Have clinically relevant hematologic, hepatic, cardiac, or renal disease.
8. Have a medical history of infection with human immunodeficiency virus, hepatitis C and/or hepatitis B, or found to have an abnormality at Screening.
9. Have a history of substance abuse (based on DSMIV criteria) within the past 12 months prior to Screening.
10. If female are pregnant or breastfeeding.
11. Have a known allergy to any ingredient in the study drug.
12. Have a history of malignancy of any type within 2 years prior to Screening. A history of surgically excised non-melanoma skin cancers, and superficial bladder or prostate cancer is permitted.
13. Have a clinically significant medical, surgical, laboratory, or behavioral abnormality which in the judgment of the site Investigator makes the subject unsuitable for the study.
14. Have any significant findings not related to HD on the screening MRI which in the judgment of the site Investigator makes the subject unsuitable for the study.
15. Have any of the following conditions (which would exclude MRI participation):

    1. An implant/device/condition that is contraindicated for MRI (e.g. pacemaker, severe claustrophobia, prosthetic heart valve, any metal fragments in the eyes or body--in some cases, an X-ray may be needed before an MRI scan, to ensure it is safe to enter the scanner).
    2. Body habitus that would impede completion of MRI scan. (Subject weight above 158 kg should be discussed with the Medical Monitor).

    NOTE: If PET is done on PET-MRI all the above conditions apply for PET-MRI.
16. Are undergoing FDG-PET and have received research-related radiation exposure that exceeds institutional guidelines in the prior year if applicable.
17. Are undergoing a LP for CSF collection and have any of the following conditions: uncorrected bleeding or clotting disorders, skin infections near the site of the LP, suspicion of increased intracranial pressure, allergies to numbing medications (local anesthetics), acute spinal trauma, history of migraines.
18. Are undergoing a LP for CSF collection and taking any of the following types of anticoagulants: coumarins and indandiones, Factor Xa inhibitors, heparins, or thrombin inhibitors.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2015-07; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Revisions to SAP were made prior to un-blinding, on June 30, 2020, upon consultation with FDA. | Prior to DBL/Study Completion
  If primary outcome, listed below (Outcome 3), does not reach its critical p-value, the secondary outcomes will not be formally tested. If both co-primary outcomes are statistically significant, the five secondary outcomes will be formally tested following a hierarchical testing procedure.
Safety and tolerability of monthly intravenous (IV) administration of pepinemab relative to placebo in subjects with early HD (Cohort B pooled, includes Cohort B1 Early Manifest and Cohort B2 Late Prodromal HD). | Up to 18 months
  Measured by drug related adverse event frequency and laboratory test abnormalities in all subjects.
Efficacy of monthly IV administration of pepinemab relative to placebo in Early Manifest HD (Cohort B1) | Up to 18 months
  Co-primary outcome measured by the change from baseline in the Huntington's Disease Two-item Cognitive Family (PTAP and OTS) selected from the Huntington's Disease

SECONDARY OUTCOMES:
Clinical feature of Early Manifest HD: motor function (Q-Motor) | Up to 18 months
  Measured by change from baseline of Q-Motor Tap Speed IOI duration mean in Cohort B1
Clinical feature of Early Manifest HD: functional capacity (UHDRS-TFC) | Up to 18 months
  Measured by change from baseline of UHDRS-TFC score in Cohort B1
Clinical feature of Early HD: functional capacity (UHDRS-TFC) | Up to 18 months
  Measured by time to 1-point change in UHDRS-TFC score in Cohort B pooled
Clinical Feature of Early HD: motor function (Q-Motor) | Up to 18 months
  Measured by change from baseline of Q-Motor Tap Speed IOI duration mean in Cohort B pooled
Clinical Feature of Early HD: cognition (Huntington's Disease Two-item Cognitive Family). | Up to 18 months
  Measured by change from baseline in the two-item HD-CAB family (PTAP and OTS) in Cohort B pooled

OTHER OUTCOMES:
Clinical feature of HD: cognition | Up to 18 months
  Measured by change from baseline in the HD-CAB composite score
Impact of monthly IV administration of pepinemab relative to placebo on change in brain metabolic activity | Up to 18 months
  Measured by change from baseline [18F]-Fluoro-2-Deoxy-D-Glucose positron emission tomography (FDG-PET) standardized uptake value ratio (SUVR) Cortical Composite Index averaging results over the right and left sides of the brain in a subset of both late prodromal and early manifest subjects
Impact of monthly IV administration of pepinemab relative to placebo on change in brain volume | Up to 18 months
  Measured by change from baseline in volumetric magnetic resonance imaging (MRI) averaging results over the right and left sides of the brain (BBSI, CBSI, VBSI, and change in white matter)
Brain metabolic activity | Up to 18 months
  Measured by change from baseline in [11C]-PBR28 translocator protein positron emission tomography (TSPO-PET) in a small subset of late prodromal subjects (Cohort B2)
pepinemab and total sSEMA4D levels in cerebral spinal fluid (CSF) | Up to 18 months
  PK parameter
Immunogenicity of monthly IV administration of pepinemab relative to placebo | Up to 18 months
  Measured by the frequency and titer of anti-drug antibodies and human anti-human antibodies
Immunophenotyping of monthly IV administration of pepinemab relative to placebo | Up to 18 months
  Measured by the levels of peripheral immune subsets in whole blood, including such lymphocyte subsets as B cells, T cells, and NK cells
Peak serum concentration (Cmax) of monthly IV administration of pepinemab | Up to 18 months
  PK parameter
Area under the serum concentration versus time curve (AUC) of monthly IV administration of pepinemab | Up to 18 months
  PK parameter
Half-life of VX15/2503 of monthly IV administration of pepinemab | Up to 18 months
  PK parameter
SEMA4D saturation in whole blood of monthly IV administration of pepinemab | Up to 18 months
  PD parameter to determine T-cell receptor occupancy
T-cell SEMA4D levels in whole blood of monthly IV administration of pepinemab | Up to 18 months
  PD parameter
Total soluble SEMA4D levels in serum of monthly IV administration of pepinemab | Up to 18 months
  PD parameter to determine the levels of total soluble SEMA4D
Clinical feature of HD: functional abilities | Up to 18 months
  Measured by change from baseline in UHDRS core functional assessments
Clinical Feature of HD: Patient Reported Outcome | Up to 18 months
  Measured by the overall response to therapy using patient reported impression of change (PGIC)
Clinical feature of HD: behavior | Up to 18 months
  Measured by change from baseline in the Problem Behavioral Assessment-Short (PBA) questionnaire
Clinical feature of HD: Patient Reported Outcome | Up to 18 months
  Measured by change from baseline in the Huntington Disease Health Index (HD-HI) Index
Clinical Safety and Non-Safety Laboratory Assessments (Clinical, Imaging, PK, PD and/or Immunogenicity) | Up to 36 months
  Dataset analysis

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Feigin, MD, Principal Investigator — The Marlene & Paolo Fresco Institute for Parkinson's & Movement Disorders-NYU Langone Medical Center
Locations (31):
- United States (28):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, San Diego, La Jolla, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado - Denver, Aurora, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - University of Florida Gainesville, Gainesville, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Columbia University, New York, New York
  - University of Rochester, Rochester, New York
  - Duke University Health Center, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Toledo, Toledo, Ohio
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Houston Medical School, Houston, Texas
  - University of Vermont, Burlington, Vermont
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington and VA Puget Sound Health Care System, Seattle, Washington
  - University of Washington, Seattle, Washington
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec

REFERENCES:
- [Background] Southwell AL, Franciosi S, Villanueva EB, Xie Y, Winter LA, Veeraraghavan J, Jonason A, Felczak B, Zhang W, Kovalik V, Waltl S, Hall G, Pouladi MA, Smith ES, Bowers WJ, Zauderer M, Hayden MR. Anti-semaphorin 4D immunotherapy ameliorates neuropathology and some cognitive impairment in the YAC128 mouse model of Huntington disease. Neurobiol Dis. 2015 Apr;76:46-56. doi: 10.1016/j.nbd.2015.01.002. Epub 2015 Feb 3. PMID 25662335
- [Derived] Estevez-Fraga C, Tabrizi SJ, Wild EJ. Huntington's Disease Clinical Trials Corner: November 2022. J Huntingtons Dis. 2022;11(4):351-367. doi: 10.3233/JHD-229006. PMID 36463457
- [Derived] Feigin A, Evans EE, Fisher TL, Leonard JE, Smith ES, Reader A, Mishra V, Manber R, Walters KA, Kowarski L, Oakes D, Siemers E, Kieburtz KD, Zauderer M; Huntington Study Group SIGNAL investigators. Pepinemab antibody blockade of SEMA4D in early Huntington's disease: a randomized, placebo-controlled, phase 2 trial. Nat Med. 2022 Oct;28(10):2183-2193. doi: 10.1038/s41591-022-01919-8. Epub 2022 Aug 8. PMID 35941373
- [Derived] Rodrigues FB, Wild EJ. Huntington's Disease Clinical Trials Corner: August 2018. J Huntingtons Dis. 2018;7(3):279-286. doi: 10.3233/JHD-189003. PMID 30103342
- See also: Nonclinical research article: Anti-semaphorin 4D immunotherapy ameliorates neuropathology and some cognitive impairment in the YAC128 mouse model of Huntington disease. — http://www.ncbi.nlm.nih.gov/pubmed/25662335